CLINICAL TRIAL: NCT01430676
Title: Risk Factors for Morbidity After Incisional Hernia Repairs
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD., Zealand University Hospital
Other Study IDs: FH-2
Record Dates: First submitted 2011-09-05; First posted 2011-09-08 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; recurrence; longterm
MeSH Terms: conditions — Incisional Hernia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Danish Ventral Hernia Database: Patients registered in the Danish Ventral Hernia Database during January 1st 2007 to december 31st 2010
  Interventions: Procedure: differences in surgical techniques

INTERVENTIONS:
Procedure: differences in surgical techniques — follow the risk for morbidity after incisional hernia repair

SUMMARY:
The Danish Ventral Hernia Database (DVHD) registers 37 different perioperative parameters. The aim of present study is to use large-scale data from DVHD to uncover risk factors for readmission, reoperation (any indication), death and reoperation for recurrence after incisional hernia repair.

DETAILED DESCRIPTION:
All principal incisional hernias registered in the Danish Ventral Hernia Database are included in the study. The included patients will be followed in up to 4 years in order to identify correlation between technical aspects of the hernia repair and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Incisional hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All incisional hernia repairs registered in tha Danish National Hernia Database from January 1st 2007 to December 31st 2010
Sampling Method: Non-Probability Sample
Enrollment: 3460 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Recurrence repair | up to 4 years
  Risk factors for recurrence repair after incisional hernia repair
Readmission | 30 days after operation
  Riskfactors for readmission within 30 days after incisional hernia repair
Reoperation | 30 days
  Riskfactors for reoperation (any procedure) within 30 days after incisional hernia repair
Death | 30 days
  Riskfactors for death within 30 days after incisional hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — dept. surgery, Køge sygehus, Denmark
Locations (1):
- Køge Hospital, Køge, Denmark